CLINICAL TRIAL: NCT03732196
Title: Reproducibility and Relative Validity of a Semi-quantitative Food Frequency Questionnaire for Chinese Pregnant Women in Hong Kong
Brief Title: Food Frequency Questionnaire for Chinese Pregnant Women
Status: Terminated | Type: Observational
Why Stopped: Unable to recruit enough participants
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ruth Chan, Senior Research Fellow, Chinese University of Hong Kong
Other Study IDs: 2018.440
Record Dates: First submitted 2018-11-01; First posted 2018-11-06 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Dietary Intake

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study aims to evaluate the reproducibility and relative validity of a semi-quantitative food frequency questionnaire (FFQ) to assess food group consumption and nutrient intake for Chinese pregnant women in Hong Kong.

A total of 100 apparently healthy pregnant women aged 18 or above and with gestational age of at least 5 weeks willl be recruited from the antenatal clinic of the Prince of Wales Hospital. The research staff will check for eligible subjects, explain study details and invite them to join the study. Written consent will be obtained from all subjects. Various maternal data will be collected using standardized methods and questionnaires, and retrieved from the hospital record.

Each participant will be asked to complete the FFQ twice within 3 to 4 weeks interval (for reproducibility evaluation), and three 24-hour food recalls in between the two administrations of the FFQ as a reference method to validate the FFQ (for validity evaluation). The three 24-hour food recalls will include two weekdays and one weekend day. On the interview day in which the 1st FFQ is administrated (FFQ1), each participant will be explained by trained research staff on how to complete the FFQ by herself with the provision of the food portion booklet. Each participant will be asked to complete the 1st FFQ regarding her intake of various food groups over the past month. The frequency of food group intake will be reported per day, week or month, and portions will be reported based on standard referent portion sizes, as pieces, glasses, cups, spoons, centilitres or grams. Data on use of supplements will be collected by asking subjects to specify the brand, the frequency, and the dosage of supplements used. On the same interview day, participant will also be asked by trained research staff to recall all foods and beverages that have been consumed over the past 24 hours. Food photo albums and eating utensils of standardized portions will be displayed to help recall. The 2nd administration of the FFQ (FFQ2) will be done 3 to 4 weeks after the 1st administration of the FFQ. The FFQ2 and the food portion booklet as well as the additional 24-hour recall forms will be given to the participants by email or post within 3 to 4 weeks after the 1st administration of the FFQ (FFQ1). Between the intervals of two FFQs, the research staff will give phone call to the participant on two separate days to complete two more 24-hour food recalls for validity evaluation purpose. Daily dietary and nutrient intake collected by both FFQs and 24-hour recalls will be entered and calculated using the nutrition analysis software Food Processor Nutrition analysis and Fitness software version 8.0 (ESHA Research, Salem, USA) including local foods selected from food composition tables from China and Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Should be Hong Kong Chinese citizen
* Should reside normally in Hong Kong
* Age at or above 18 years old
* With antenatal registry in the study hospital
* Singleton pregnancy
* Gestational age of 5 weeks or above
* Could speak and understand Chinese
* Willing to follow the study procedures

Exclusion Criteria:

* Currently participating in any clinical trial or trial with dietary intervention
* Multiple pregnancy
* With any renal, liver or thyroid dysfunction, any other indication of a major medical or psychological illness, as judged by the investigators as ineligible to participate the study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: A total of 100 apparently healthy pregnant women aged 18 or above and with gestational age of at least 5 weeks willl be recruited from the antenatal clinic of the Prince of Wales Hospital. The research staff will check for eligible subjects, explain study details and invite them to join the study. Written consent will be obtained from all subjects. Various maternal data will be collected using standardized methods and questionnaires, and retrieved from the hospital record.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Difference in dietary intakes | Baseline
  Difference in dietary intakes measured using Food Frequency Questionnaire and multiple 24-hour recalls will be examined

SECONDARY OUTCOMES:
Change in dietary intakes | Change betwen baseline and one month
  Change in dietary intakes measured using Food Frequency Questionnaire at baseline and one month will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China